CLINICAL TRIAL: NCT04198493
Title: Impact of Continuous Positive Airway Pressure Treatment on Cognitive Function in Adults With Down Syndrome With Obstructive Sleep Apnea
Brief Title: Effect of CPAP Treatment in Cognition in Adults With DS and OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-SAH-2019-62
Record Dates: First submitted 2019-11-28; First posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Down Syndrome; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Open pilot study with randomized therapeutic intervention of parallel groups and blind evaluation in neuropsychological assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Positive Airway Pressure(CPAP) (Experimental): Patients with CPAP treatment. Titration will be performed by polysomnography CPAP to determine the optimal treatment pressure.
  This group will also be instructed in sleep hygiene and dietary counseling
  Intervention:
  Device: CPAP Other: Conservative treatment for OSA
  Interventions: Device: CPAP; Other: CONSERVATIVE TREATMENT for OSA
- CONSERVATIVE TREATMENT for OSA (Active Comparator): Sleep hygiene and dietary counseling. Sleep hygiene (regular sleep schedule, physical exercise) and dietary counseling Intervention: Other: Conservative treatment for OSA
  Interventions: Other: CONSERVATIVE TREATMENT for OSA

INTERVENTIONS:
Device: CPAP — CPAP treatment every night plus conservative treatment for OSA: sleep hygiene and dietary counseling
  Arms: Continuous Positive Airway Pressure(CPAP)
Other: CONSERVATIVE TREATMENT for OSA — Conservative treatment for OSA: sleep hygiene and dietary counseling

SUMMARY:
Adults with Down syndrome (DS) have a high prevalence of obstructive sleep apnea (OSA), which may worsen cognitive performance.

In general population, continuous positive airway pressure (CPAP), the gold Standard treatment for OSA, partially reverses cognitive impairment secondary to OSA. CPAP treatment, however, is not regularly proposed in adults with DS and OSA. It is usually presumed both by caregivers and physicians, that DS patients will not tolerate or adapt to the treatment, and that they would not benefit much more from CPAP treatment. Therefore, data about the feasibility and impact of CPAP treatment on cognitive function in this population is lacking.

The main objective of this study is to investigate cognitive performance in adults with DS and OSA, the corresponding functional brain changes and their reversibility with CPAP treatment.

DETAILED DESCRIPTION:
Population Participants will be included from the Catalan Down Syndrome Foundation (FCSD). After obtaining a written informed consent, approved by the ethical committee, a total of 60 adult subjects of both sexes with SD and without dementia will be included. Forty subjects with a diagnosis of severe OSA (AHI> 30) without significant comorbidities or excessive daytime sleepiness (Epworth <12) and 20 subjects without OSA.

Objectives:

The general objective is to evaluate cognitive and/or behavioural dysfunction in adults with Down syndrome that can improve with CPAP treatment.

* By evaluating sleep, cognitive function and behaviour aspects in adults with Down syndrome with and without OSA.
* By assessing the changes in sleep, in cognitive, behavioural function, and brain connectivity measures after 6 month of treatment in subjects with DS and severe OSA.

Secondary objectives:

* Assess the relationship between the severity of OSA (AHI, hypoxemia, sleep fragmentation) and severity in cognitive impairment.
* Identify possible sleep and anthropometric parameters that could suggest a worsening in cognitive function in subjects with DS and OSA.

Methodology:

Open pilot study with randomized therapeutic intervention of parallel groups and blind evaluation in neuropsychological assessment.

Patients with severe OSA will be randomized to i) conservative treatment (CT) or to ii) CPAP and conservative treatment.

Patients included in the study will be monitored and followed for 6 months. Patients with severe OSA will perform follow up visits to monitor the objective compliance and side effects of the treatment in the 1st, 3rd and 6th month.

At baseline and after 6 months of treatment, in the three groups of subjects (i) Subjects without OSA, ii) Subjects with OSA and CPAP treatment, and iii) Subjects with OSA+ TC treatment , it will be performed:

1. Sleep evaluation:

   Subjective sleep quality (Pittsburgh sleep quality index) and daytime Somnolence (Epworth Sleepiness Scale) Nocturnal sleep by polysomnography (PSG) Sleep-wake pattern by actigraphy
2. Neurocognitive function with an extensive neuropsychological battery assessing mainly memory, attention and executive functions for DS population. (CAMCOG-DS, Cued Recall Test (CRT), different subtests of the Barcelona Test battery: orientation in person, time and space, language items (comprehension, reading and writing), verbal abstraction and oculomotor praxis, cats and dogs test, Attention cancellation test, verbal fluency test.
3. Measures of cerebral functional connectivity: through measures of consistency, mutual information, probability of synchronization and transfer entropy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes with ages over 18 years old with DS.
* A good general health with adequate visual and auditory acuity will be required
* Understanding and accepting the study procedures and signing an informed consent (guardian and / or patient).
* intelligence quotient(IQ) ratio> 34 (mild and moderate severe intellectual disability according to the International Statistical Classification of Diseases and Related Health Problems, ICD-10, criteria).
* Subjects without dementia: Absence of loss of cognitive functions (demonstrated by the longitudinal administration of neuropsychological tests and verified by family members)
* Absence of psychiatric comorbidity

Exclusion Criteria:

* Severe intellectual disability (due to limitations in cognitive tests)
* Presence of psychiatric pathology, unstable disease, cardiac or respiratory failure.
* Intake of psychoactive drugs in the three months prior to the study.
* Patients diagnosed with OSA, undergoing treatment with CPAP.
* Subjects with an Epworth Sleep Scale score > 12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of the changes on cognitive attentional tasks | Baseline and after 6 months of treatment
  psychomotor speed (in seconds) performing an attentional task
Changes in cerebral functional connectivity | Baseline and after 6 months of treatment
  Significant probability maps (SPM) showing statistical changes on connectivity measures between sleep stages

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Sleep Unit. Hospital de la Santa Creu i Sant Pau, Barcelona, Spain